CLINICAL TRIAL: NCT03528330
Title: Clinical, Radiological and Microbiological Outcomes of Implants With Two Different Connection Configurations, a Split-mouth RCT.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Assistanat Postdoctoral Lecturer (Profesor Ayudante Doctor), University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H1506438439563
Record Dates: First submitted 2018-03-03; First posted 2018-05-17 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Bone Loss, Alveolar; Dental Implant Failed
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Rehabilitation; Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal hexagon connection (Active Comparator): Small flaps will be elevated to reduce any kind of injury on the periosteum and maintain the blood supply during the healing period.
  Patients will receive 2 implants. One implant (assigned randomly) will have internal hexagon connection.
  The Internal Hex (IH) implant has a 2.5mm internal hexagon and a 90° cone. The platform diameter is Ø3.5mm.
  Interventions: Device: Rehabilitation with dental implant with internal hexagon connection
- Conical connection (Experimental): Small flaps will be elevated to reduce any kind of injury on the periosteum and maintain the blood supply during the healing period.
  Patients will receive 2 implants. One implant (assigned randomly) will have internal hexagon connection.
  The Conical Standard (CS) implant has a 2.5mm internal hexagon and 22° cone. The platform diameter is Ø3.1mm.
  Interventions: Device: Rehabilitation with dental implant with conical connection

INTERVENTIONS:
Device: Rehabilitation with dental implant with internal hexagon connection — All patients will receive an implant with internal hexagon connection. All implants will be10 mm in length and 3.75 mm in diameter. Implants will be inserted slightly subcrestal. Bone levels will be measured using a calibrated probe.
  Torque insertion will be assed using W&H machine Once inserted, implants will be connected to smart pegs to test primary stability.
  A periapical x-ray will be done after the operation. Thereafter, a specific coping for digital impression will be connected to the implant and a digital impression will be taken. Aim of this procedure will be to produce a screw retained definitive zirconia prosthesis to be adapted at the time of second surgery
  Arms: Internal hexagon connection
Device: Rehabilitation with dental implant with conical connection — All patients will receive an implant with conical connection. All implants will be10 mm in length and 3.75 mm in diameter. Implants will be inserted slightly subcrestal. Bone levels will be measured using a calibrated probe.
  Torque insertion will be assed using W&H machine Once inserted, implants will be connected to smart pegs to test primary stability.
  A periapical x-ray will be done after the operation. Thereafter, a specific coping for digital impression will be connected to the implant and a digital impression will be taken. Aim of this procedure will be to produce a screw retained definitive zirconia prosthesis to be adapted at the time of second surgery
  Arms: Conical connection

SUMMARY:
This study designed as a randomized controlled split-mouth trial will be conducted at the Dental Clinic of the University of Valencia. The aim will be to assess differences in clinical, radiological and microbiological outcomes between implants with 2 different connections: internal hexagon and conical connection. Following the premises, to minimize the bias related to prosthetic phase and maximize the effect of connections on MBL changes, a 1abutment-1time protocol will be used.

The study hypothesis is that there will be no statistically significant differences between both implant connections.

ELIGIBILITY:
Inclusion Criteria:

* able to sign an informed consent form
* aged 25 years or more
* Any patient requiring two implant-supported crowns in the lower or upper jaw
* Kennedy class I, II, and III;
* teeth extracted at least 6 months before implant placement;
* sufficient bone volumes to accommodate dental implants without augmentation procedure

Exclusion Criteria:

* General medical and/or psychiatric contraindications to implant surgery,
* Pregnancy or nursing,
* Heavy smoking (more than 10 cigarettes/day),
* Treatment with anticoagulant drugs (International Normalized Ratio under 1.8), bisphosphonates, steroid therapy or anticonvulsants drugs.
* No regenerated bone
* Untreated Periodontal disease and inability of the patient to maintain reasonable oral hygiene according to study requirements.
* Patients with history of alcohol, narcotics or drug abuse. (Alcoholism: more than two bottles of beer per day)
* Patients receiving radiotherapy, chemotherapy or any other immunosuppressive treatment, or who have been administered radiotherapy in the last 5 years. (Patients through at any time received radiotherapy to the head and neck region should be excluded anyway.)
* Metabolic bone disorders
* Uncontrolled bleeding disorders such as: hemophilia, thrombocytopenia, granulocytopenia.
* Degenerative diseases.
* Osteoradionecrosis.
* Renal failure.
* Organ transplant recipients.
* HIV positive.
* Malignant diseases.
* Diseases that compromise the immune system.
* Unbalanced diabetes mellitus. (HbA1c above 6.5), Uncontrolled endocrine diseases
* Psychotic diseases.
* Hypersensitivity to one of the components of the implant in general and titanium in particular.
* Women who are pregnant or lactating.
* Lack of patient cooperation.
* Parafunctional habits, such as Bruxism or Temporomandibular joint disease.
* Various pathologies of the oral mucosa for example: Benign mucous pemphigoid, desquamative ginigivitis, erosive lichen planus, malignancy of oral cavity, bolus erosive diseases of the oral mucosa.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Peri-implant bone level changes | a. implant placement (baseline), b. abutment connection (8-12 weeks), c. after 1 year of function (14-15 months), d. after 3 years of function (38-39 months).
  calculated using intraoral digital periapical radiographs

SECONDARY OUTCOMES:
Implant failure | 3 years
  Requiring removal
Prosthetic complications | 3 years
  Screw loosening or fracture, fracture of the prosthesis or of the ceramic
Resonance frequency analysis values | a. implant placement (baseline) b. abutment connection (8-12 weeks)
  Measured using Ostell Mentor
Probing pocket depth | a. implant placement (baseline), b. abutment connection (8-12 weeks), c. after 1 year of function (14-15 months), d. after 3 years of function (38-39 months).
  Measurement of peri-implant pocket depth with a periodontal probe
Microbial loads | 12 months after loading
  Quantities of different microbial species assessed using 16s metagenomics
Plaque | a. implant placement (baseline), b. abutment connection (8-12 weeks), c. after 1 year of function (14-15 months), d. after 3 years of function (38-39 months).
  Presence or absence of plaque
Bleeding on probing | a. implant placement (baseline), b. abutment connection (8-12 weeks), c. after 1 year of function (14-15 months), d. after 3 years of function (38-39 months).
  Presence or absence of bleeding after probing pocket depth

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Odontológica de la Universitat de Valencia, Fundación Lluis Alcanyis, Valencia, Spain